CLINICAL TRIAL: NCT06727136
Title: A Phase 1, Open-label Study to Characterize Single and Repeat Dose Pharmacokinetics (Including Food Effect) of Tebipenem-pivoxil-hydrobromide and Its Major Metabolite (SPR1349) in Healthy Participants
Brief Title: A Study to Characterize Single and Repeat Dose Pharmacokinetics of Tebipenem-Pivoxil-Hydrobromide (TBP-PI-HBr) and Its Major Metabolite (SPR1349) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPR994-110
Record Dates: First submitted 2024-12-06; First posted 2024-12-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — tebipenem

STUDY DESIGN:
Intervention Model Description: The study involves 2 parts (A and B) and 3 cohorts (Cohort 1, 2 and 3) of which Cohort 2 has a crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Cohort 1 (Experimental): Participants will receive TBP-PI-HBr, 900 milligrams (mg) tablets orally, as a single dose under fasted condition on Day 1.
  Interventions: Drug: TBP-PI-HBr
- Part A: Cohort 2 (Fasted/Fed) (Experimental): Participants will receive TBP-PI-HBr, 1200 mg, tablets, orally, as a single dose under fasted and fed conditions on Day 1 and Day 3, as per the assigned crossover sequence.
  Interventions: Drug: TBP-PI-HBr
- Part B: Cohort 3 (Experimental): Participants will receive TBP-PI-HBr, 600 mg, orally as a single dose on Day 1, followed by 9 doses every 6 hours from Day 3 through Day 5. (first and ninth dose will be given under fasted conditions).
  Interventions: Drug: TBP-PI-HBr

INTERVENTIONS:
Drug: TBP-PI-HBr — TBP-PI-HBr film-coated immediate-release tablets
  Other Names: SPR994

SUMMARY:
The main purpose of the study is to characterize the systemic pharmacokinetic (PK) parameters (plasma, whole blood) of tebipenem (TBP) pharmacologically active moiety of tebipenem-pivoxil-hydrobromide (TBP-PI-HBr) and its urinary excretion at different dose levels in healthy participants. The study also aims to assess the plasma and urine PK parameters of SPR1349, a major metabolite of TBP.

ELIGIBILITY:
Inclusion Criteria

* Participants who are healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG).
* Body weight considering body mass index (BMI) within the range of 18 to 32 kilogram per meter square (kg/m^2), inclusive.
* Participant must be 18 (or the legal age of consent in the jurisdiction in which the study is taking place) to 55 years of age inclusive, at the time of signing the informed consent.

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular (CV), respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or study procedures or interfering with the interpretation of data.
* Past or intended use of over-the-counter or prescription medication including herbal medications within 28 days prior to dosing, with the exception of supplemental vitamins, hormonal medications (contraceptives or hormone-replacement therapy), or occasional oral acetaminophen (not to exceeding 2 g total daily dose).
* Current enrollment or past participation in another investigational/observational clinical study in which an investigational intervention (e.g., drug, vaccine, invasive device) was administered within the last 30 days, or 5 half-lives whichever is longer.
* Positive COVID-19 screening test using PCR or antigen assay at Day -1
* Donation of, or significant blood loss of, more than 500 mL of blood within 56 days prior to dosing.
* Receipt of a blood transfusion within 1 year prior to enrollment or plasma donation within 7 days prior to dosing.
* QTc >450 msec.

Note: Other inclusion/exclusion criteria may also apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
Part A and B: Maximum Observed Concentration (Cmax) of TBP in Plasma and Blood | Cohort 1: Pre-dose and at multiple timepoints post-dose up to Day 3; Cohort 2: Pre-dose and at multiple timepoints post-dose up to Day 5; Cohort 3: pre-dose and at multiple timepoints post-dose up to Day 7
Part A and B: Time to Cmax (Tmax) of TBP in Plasma and Blood | Cohort 1: Pre-dose and at multiple timepoints post-dose up to Day 3; Cohort 2: Pre-dose and at multiple timepoints post-dose up to Day 5; Cohort 3: pre-dose and at multiple timepoints post-dose up to Day 7
Part A and B: Area Under the Concentration-Time Curve (AUC) Extrapolated to Infinity [AUC(0-inf)] of TBP in Plasma and Blood | Cohort 1: Pre-dose and at multiple timepoints post-dose up to Day 3; Cohort 2: Pre-dose and at multiple timepoints post-dose up to Day 5; Cohort 3: pre-dose and at multiple timepoints post-dose up to Day 7
Part A and B: AUC From Time Zero to the Time of the Last Evaluable Concentration [AUC(0-t)] of TBP in Plasma and Blood | Cohort 1: Pre-dose and at multiple timepoints post-dose up to Day 3; Cohort 2: Pre-dose and at multiple timepoints post-dose up to Day 5; Cohort 3: pre-dose and at multiple timepoints post-dose up to Day 7
Part A and B: Amount Excreted in Urine (Ae) of TBP | Cohort 1: Pre-dose and at multiple timepoints post-dose up to Day 3; Cohort 2: Pre-dose and at multiple timepoints post-dose up to Day 5; Cohort 3: pre-dose and at multiple timepoints post-dose up to Day 7
Part A and B: Fraction of Dose Excreted in Urine (Fe) of TBP | Cohort 1: Pre-dose and at multiple timepoints post-dose up to Day 3; Cohort 2: Pre-dose and at multiple timepoints post-dose up to Day 5; Cohort 3: pre-dose and at multiple timepoints post-dose up to Day 7
Part B: AUC From Time Zero to 6 Hours Post-dose AUC(0-6) of TBP in Plasma and Blood | Pre-dose and at multiple timepoints post-dose up to Day 7
Part B: Ae of SPR1349 | Pre-dose and at multiple timepoints post-dose up to Day 7
Part B: Fe of SPR1349 | Pre-dose and at multiple timepoints post-dose up to Day 7

SECONDARY OUTCOMES:
Part B: Tmax of SPR1349 in Plasma | Pre-dose and at multiple timepoints post-dose up to Day 7
Part B: Cmax of SPR1349 in Plasma | Pre-dose and at multiple timepoints post-dose up to Day 7
Part B: AUC(0-inf) of SPR1349 in Plasma | Pre-dose and at multiple timepoints post-dose up to Day 7
Part B: AUC(0-t) of SPR1349 in Plasma | Pre-dose and at multiple timepoints post-dose up to Day 7
Part B: AUC(0-6) of SPR1349 in Plasma | Pre-dose and at multiple timepoints post-dose up to Day 7
Part B: Plasma AUC Ratio of SPR1349 to TBP | Pre-dose and at multiple timepoints post-dose up to Day 7
Part B: Ae Ratio of SPR1349 to TBP | Pre-dose and at multiple timepoints post-dose up to Day 7
Parts A and B: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 to Day 21

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Facility, Salt Lake City, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No